CLINICAL TRIAL: NCT05001399
Title: Feasibility of Using Holographic Memory Resolution® (HMR) in Patients/Clients With Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Billings Clinic (Other)
Collaborators: Healing Dimensions, ACC (Unknown)
Responsible Party: Principal Investigator, Mary Gaddy, Prinicipal Investigator, Billings Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21.012
Record Dates: First submitted 2021-07-29; First posted 2021-08-12 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Chronic Pain; Headache, Migraine; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Chronic Pain; Migraine Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Pilot and Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Holographic Memory Resolution® (HMR) Intervention (Experimental): Intervention will be comprised of 4 sessions lasting approximately 90 minutes at one of two sites, Billings Clinic in Billings, Montana or Healing Dimensions AAC in Tucson, Arizona. The 4 sessions will be completed in approximately 9 weeks.
  Interventions: Behavioral: Holographic Memory Resolution® (HMR)

INTERVENTIONS:
Behavioral: Holographic Memory Resolution® (HMR) — Clients will participate in Holographic Memory Resolution® (HMR) administered by a trained HMR practitioner. Clients will be introduced to relaxation techniques and safe scene identification. This exercise encourages the client to identify a place in which they feel safe and where nobody can be there without client's invitation. Clients will then describe the place and associated colors of the experience, how the colors move in their body, and how they move through their safe scene. The subsequent 2-3 sessions will continue to explore safe scene and color therapy.

SUMMARY:
Study Purpose: This study will explore the feasibility of administering Holographic Memory Resolution® (HMR) to adults who are experiencing chronic pain for 6 months or more.

DETAILED DESCRIPTION:
Chronic pain is a significant health care problem and is one of the most common reasons individuals seek medical care. It is estimated that approximately 20.4% (50 million) of U.S. adults suffer from chronic pain, and 8% of those adults consider the pain to have high-impact on their quality of life. Chronic pain is also linked to many physical and mental health conditions, and for the most part, effective and safe strategies are lacking. While opioids are an option in the management of chronic pain, opioid misuse and abuse is common, making this a less desirable strategy. As noted, mental health concerns often co-exist with chronic pain. Depression and mental health concerns are skyrocketing across the U.S. Nearly one in five U.S. adults live with a mental illness, and only 50% of people with mental illnesses receive treatment. For those who do receive treatment, symptom resolution can be incomplete, and some psychotropic medications induce unwanted side effects, leading to decreased adherence and withdrawal of care.

Due to the scarcity of effective interventions to manage both chronic pain and mental health disorders, mind body interventions (MBI) are sometimes employed in these individuals. MBI are defined as a variety of activities that exercise and encourage mental and/or physical fitness. Lists of MBIs include diverse activities such as yoga, meditation, hypnosis, dance, or music therapy. Past meta-analyses have noted that primary studies on effective MBI to manage conditions such as fibromyalgia and depression in chronic pain are lacking. More recent publications indicate this is no longer the case. MBI may demonstrate small to moderate effects sizes in some populations for at least a short amount of time.

Holographic Memory Resolution® (HMR) is a proposed MBI for this study. HMR was developed by Brent Baum in the early 1990's, and he and several others have been using the technique to treat individuals with a variety of complaints including depression, anxiety, pain, post-traumatic stress disorder and related conditions. HMR incorporates elements of energy psychology, Eastern philosophical tradition, hypnosis, guided imagery, and clean-language interviewing into a single approach with the aim of changing the emotional component of a negative memory to resolve psychological distress. Despite being used for several decades, HMR appears to have received little attention in scientific literature. Only one citation appears in the National Library of Medicine, and this author only describes the technique. Theoretical, qualitative and quantitative studies of HMR appear to be non-existent in peer-reviewed literature.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years or older
* Suffering from pain of 4 or greater intensity on a 0-10 scale with "0" being no pain and "10" being worst possible pain.
* Pain symptoms will have been present for at least 6 months. Patients with chronic migraine headaches will be eligible if headaches occur at least every two months.
* Associated symptoms could include anxiety, depression, or physical symptoms such as pain, migraines, or other symptoms that have interfered with quality of life or work/life balance.
* Interested clients will have primary care provider agreement to participate in the study.

Exclusion Criteria:

* Diagnosis of psychosis or schizoaffective disorder, personality disorder, or suicidal ideation.
* Clients taking mood altering substances and those that have a propensity toward altering delta, theta, alpha, and beta wave ranges will be excluded. These substances include but are not limited to Cannabis/Marijuana/ hashish/THC, PCP, phencyclidine, or Angel dust, Barbiturates, Benzodiazepines, Opioids/heroin, Clozapine (+++delta/slow waves/- - alpha waves), Lithium, Stimulants/ (Illicit: Cocaine, Methamphetamine), and Hallucinogens/MDMA (ecstasy)/LSD.
* Clients who ingest alcohol must be 3 months abstinent/in recovery before session if alcohol dependent and 48 hours abstinent before session if not alcohol dependent/in recovery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Completion Rate of an HMR Intervention | Following 4 HMR sessions, approximately 8-9 weeks per participant.
  The percentage of patients who complete 4 HMR sessions.

SECONDARY OUTCOMES:
Somatic Symptomatic Scale (SSS-8) | Baseline, prior to Session 3 ( Day 14-24), prior to Session 4 (8-9 weeks), and 1 month after Session 4.
  The SSS-8, an abbreviated version of the PHQ-15, is a validated 8-item client-report measure of somatic symptom burden. Respondents are asked to answer the question "During the past 7 days, how much have you been bothered by any of the following problems?" concerning gastrointestinal, pain, fatigue, and cardiopulmonary aspects. Items are scored on a 5-point Likert scale (0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, 4=Very much). Somatic symptom scoring ranges from 0-32 [(no to minimal (0-3 points), low (4-7 points), medium (8-11 points), high (12-15 points), and very high (16-32 points)].

CONTACTS AND LOCATIONS:
Overall Officials: Mary Gaddy, MD, Principal Investigator — Billings Clinic
Locations (2):
- United States (2):
  - Healing Dimensions ACC, Tucson, Arizona
  - Billings Clinic, Billings, Montana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahlhamer J, Lucas J, Zelaya C, Nahin R, Mackey S, DeBar L, Kerns R, Von Korff M, Porter L, Helmick C. Prevalence of Chronic Pain and High-Impact Chronic Pain Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Sep 14;67(36):1001-1006. doi: 10.15585/mmwr.mm6736a2. PMID 30212442
- [Background] Voon P, Karamouzian M, Kerr T. Chronic pain and opioid misuse: a review of reviews. Subst Abuse Treat Prev Policy. 2017 Aug 15;12(1):36. doi: 10.1186/s13011-017-0120-7. PMID 28810899
- [Background] Fava M, Judge R, Hoog SL, Nilsson ME, Koke SC. Fluoxetine versus sertraline and paroxetine in major depressive disorder: changes in weight with long-term treatment. J Clin Psychiatry. 2000 Nov;61(11):863-7. doi: 10.4088/jcp.v61n1109. PMID 11105740
- [Background] Lieberman JA, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Keefe RS, Davis SM, Davis CE, Lebowitz BD, Severe J, Hsiao JK; Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Investigators. Effectiveness of antipsychotic drugs in patients with chronic schizophrenia. N Engl J Med. 2005 Sep 22;353(12):1209-23. doi: 10.1056/NEJMoa051688. Epub 2005 Sep 19. PMID 16172203
- [Background] Theadom A, Cropley M, Smith HE, Feigin VL, McPherson K. Mind and body therapy for fibromyalgia. Cochrane Database Syst Rev. 2015 Apr 9;2015(4):CD001980. doi: 10.1002/14651858.CD001980.pub3. PMID 25856658
- [Background] Sud A, Lai KSP, Cheng DK, Chung C, Pico-Espinosa OJ, Rice DB. Mind-Body Interventions for Depressive Symptoms in Chronic Pain: A Systematic Review of Meta-Analyses. Pain Physician. 2021 Jan;24(1):61-72. PMID 33400428
- [Background] Gomez-de-Regil L, Estrella-Castillo DF. Psychotherapy for Physical Pain in Patients with Fibromyalgia: A Systematic Review. Pain Res Manag. 2020 Jul 4;2020:3408052. doi: 10.1155/2020/3408052. eCollection 2020. PMID 32714478
- [Background] Kwon CY, Lee B, Chung SY, Kim JW. Do Cochrane reviews reflect the latest evidence on meditation and mindfulness-based interventions? A snapshot of the current evidence. Explore (NY). 2021 Nov-Dec;17(6):557-565. doi: 10.1016/j.explore.2020.05.016. Epub 2020 May 30. PMID 32527685
- [Background] Brandman W. Integrative perspectives. Holographic memory resolution. Perspect Psychiatr Care. 2005 Jul-Sep;41(3):139-41. doi: 10.1111/j.1744-6163.2005.00026.x. No abstract available. PMID 16138824
- [Background] Murphy A, Steele M, Dube SR, Bate J, Bonuck K, Meissner P, Goldman H, Steele H. Adverse Childhood Experiences (ACEs) questionnaire and Adult Attachment Interview (AAI): implications for parent child relationships. Child Abuse Negl. 2014 Feb;38(2):224-33. doi: 10.1016/j.chiabu.2013.09.004. Epub 2013 Oct 24. PMID 24670331
- [Background] Gierk B, Kohlmann S, Kroenke K, Spangenberg L, Zenger M, Brahler E, Lowe B. The somatic symptom scale-8 (SSS-8): a brief measure of somatic symptom burden. JAMA Intern Med. 2014 Mar;174(3):399-407. doi: 10.1001/jamainternmed.2013.12179. PMID 24276929
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Chen B, Van Assche J, Vansteenkiste M, Soenens B, Beyers W. Does Psychological Need Satisfaction Matter When Environmental or Financial Safety are at Risk? Journal of Happiness Studies. 2015;16(3):745-766.
- [Background] Chen B, Vansteenkiste M, Beyers W, et al. Basic psychological need satisfaction, need frustration, and need strength across four cultures. Motivation and Emotion. 2015;39(2):216-236.
- [Background] Nix G, Ryan R, Manly JB, Deci E. Revitalization through Self-Regulation: The Effects of Autonomous and Controlled Motivation on Happiness and Vitality. Journal of Experimental Social Psychology. 1999;35:266-284.
- [Background] Bostic TJ, Rubio DM, Hood M. A validation of the subjective vitality scale using structural equation modeling. Social Indicators Research. 2000;52(3):313-324.
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Derived] Welsh JW, Durham RM, Sitar SI, Modisette KC, Estrada BD, Dennis ML. Diagnosing Adolescent Substance Use and Co-Occurring Disorders Using the Global Appraisal of Individual Needs Quick Version-4. Psychiatr Res Clin Pract. 2024 Jun 28;6(4):143-150. doi: 10.1176/appi.prcp.20230078. eCollection 2024 Winter. PMID 39669537
- [Derived] Gaddy MD, Baum B, Kiesow B, Coombs NC, Beamon ER, Mullowney Y, Williams GC, Brant JM. The Use of Holographic Memory Resolution(R) to Improve the Physical and Biopsychosocial Symptoms of Chronic Pain: A Feasibility, Mixed Methods Study. Psychiatr Res Clin Pract. 2023 Sep 19;6(1):4-11. doi: 10.1176/appi.prcp.20230028. eCollection 2024 Spring. PMID 38510483
- See also: National Institute of Mental Health. Mental Health Information. 2020. — http://www.nimh.nih.gov/health/topics/index.shtml